CLINICAL TRIAL: NCT03145103
Title: Clinical Safety and Efficacy of Hydrophilic Acrylic Intraocular Lenses - Retro Prospective Study
Brief Title: Clinical Safety and Efficacy of Hydrophilic Acrylic Intraocular Lenses
Acronym: UVEA409
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASPHINA 409-BER-401-17
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 409M (Experimental): CT ASPHINA 409M IOL
  Interventions: Device: CT ASPHINA 409

INTERVENTIONS:
Device: CT ASPHINA 409 — intraocular lens

SUMMARY:
Clinical safety and efficacy of CT ASPHINA 409 IOLs after implantation

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent;
* Patients of any gender
* Assured follow-up examinations
* Biometry measurement preferably compatible with the IOLMaster evaluation;
* IOL implanted into the capsular bag with IOL model CT ASPHINA 409MP (UVE material) in one eye with at least 12 months follow up at the time of the postop visit
* Patients who had uncomplicated (no peroperative complication) aged-related cataract surgery in a healthy eye (beside clinically significant cataract)

Exclusion Criteria:

* BCVA not available preoperatively or better than 0.3 logMAR pre-op
* Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial
* Patients whose freedom is impaired by administrative or legal order
* Concurrent participation in another drug or device investigation -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 to 18 months after surgery
  Monocular best corrected distance visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansson B, Daniel ACS, Herbers C, Gerl M, Kretz FTA. Clinical safety and efficacy of a hydrophilic acrylic intraocular lens in a real-world population: a 1-year follow-up retro-prospective study. BMC Ophthalmol. 2020 Jun 11;20(1):224. doi: 10.1186/s12886-020-01493-y. PMID 32527240